CLINICAL TRIAL: NCT04337021
Title: Caregiver SOS: An Intervention for Employed Caregivers
Brief Title: Caregiver Self-Management of Stress
Acronym: Caregiver SOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: The VA Western New York Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIR 18-290; 01845 (Other: CMCVAMC IRB); 2020-009 (Other: VAWNYHS IRB)
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Caregiver Distress; Job Stress
Keywords: psychological stress; family caregivers; work stress; spouse caregivers; life stress
MeSH Terms: conditions — Occupational Stress; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Caregiver SOS is delivered by phone and offers evidence-based, work and CG role performance-focused self-management counseling to employed CGs. The program includes 6, 1-hour telephonic sessions with a care manager.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caregiver SOS (Active Comparator): SOS care is brief, telephonic care (6 one-hour sessions over 3-4 months) tailored to the CG's needs, preferences, and priorities. SOS care addresses both work and caregiving-related stress. The five pillars of behavior change in SOS care are: 1) knowledge of work and CG stress; 2) stress management skills and abilities; 3) supports and resources; 4) confidence and motivation to modify stress; and 5) work and CG-focused problem-solving skills. The pillars are addressed through seven modules. In six sessions, the CM will cover each module at least once. SOS care involves an ongoing process of formulating self-management goals and action plans and preparing CGs to succeed in implementing them. Addressing both work and caregiving contexts, CMs will educate CGs about stress. CMs introduce strategies for self-managing stress and collaboratively design experiments to test these strategies. The CG's progress is monitored to identify strategies that effectively achieve self management goals.
  Interventions: Behavioral: Caregiver SOS
- Usual Care (No Intervention): CGs in this arm will be contacted telephonically once by a CM. After a brief needs assessment, the CM will provide contact information for appropriate VA (e.g., local CSP clinicians) and non-VA community resources/services. CGs will be sent brochures for the national VA CSP. Information on both the program's website (which includes links to training, education, resources, and outreach programs for CGs) and the national CG hotline number will be included in the mailed packet. After this initial contact, CGs in this group will only be contacted again 4 and 9 months after baseline for administration of follow-up research assessments. CGs will be encouraged to seek medical, psychological, social support, and social services that are available to them through VAMCs or any other non-VA/community source. CGs in the SOS group will be offered similar information.

INTERVENTIONS:
Behavioral: Caregiver SOS — SOS care is brief, telephonic care (6 one-hour sessions over 3-4 months) tailored to the CG's needs, preferences, and priorities. SOS care addresses both work and caregiving stress. The five pillars of behavior change in SOS care are: 1) knowledge of work and CG stress; 2) stress management skills and abilities; 3) supports and resources; 4) confidence and motivation to modify stress; and 5) work and CG-focused problem-solving skills. The pillars are addressed through seven modules. In six sessions, the CM will cover each module at least once. SOS care involves an ongoing process of formulating self-management goals and action plans and preparing CGs to succeed in implementing them. Addressing both work and caregiving contexts, CMs will educate CGs about stress. CMs introduce strategies for self-managing stress and collaboratively design experiments to test these strategies. The CG's progress is monitored to identify strategies that effectively achieve self management goals.
  Arms: Caregiver SOS

SUMMARY:
Unpaid informal caregivers (CGs), such as family and friends, who are also employed may be at significant risk of experiencing burden and stress. This may be especially true for CGs who provide care to care recipients coping with behavioral health issues associated with conditions like depression, anxiety, post-traumatic stress disorder and traumatic brain injury. Stress not only increases the CG's risk of workplace difficulties, illness, and poor quality of life, but also impacts the CG's ability to provide care for the care recipient. The primary aim of this randomized study is to examine the impact of a novel intervention, Caregiver SOS (Self-Management of Stress), on CG distress and work performance and productivity. Caregiver SOS is delivered by phone and offers evidence-based, work and CG role performance-focused self-management counseling to employed CGs. Study findings will ultimately shed light on whether a program that specifically addresses caregiving-work balance is effective in improving CGs' wellbeing and work functioning and the quality of Veterans' care.

DETAILED DESCRIPTION:
Background: Research has shown that unpaid, informal caregivers (CGs), such as family and friends, who are also employed may be at significant risk of experiencing burden and stress. A recent national survey found that approximately 60% of employed CGs had significant problems balancing work and caregiving. Stress not only increases the CG's risk of illness and diminishes their quality of life; it also impacts the CG's ability to provide care for the care recipient (CR) and overall relationship quality. Moreover, while work frequently adds to the CG's stress, relinquishing work can create new stress for both the CG and CR, particularly when it involves losses in resources such as income, benefits, social contacts and/or respite from caregiving duties.

Specific Aims: The aims of this study are to, 1) determine the extent to which, relative to usual care, a novel intervention providing evidence-based, telephonic CG/work stress self-management counseling is related to changes in CG psychological distress and ability to function effectively in work and CG roles, and 2) evaluate whether participation in the intervention is related to CGs' overall wellbeing and CRs' health care utilization.

Methodology: The investigators will conduct a randomized controlled trial and compare pre/post changes among 300 CGs allocated to the Caregiver SOS (for Self-Management of Stress) program or usual care. CGs who, 1) care for Veterans diagnosed with depression, anxiety, PTSD, and/or traumatic brain injury (TBI) and, 2) screen positive for clinically significant distress and CG/work role difficulty will be recruited to participate from two VA Medical Centers and their affiliated outpatient clinics. A novel intervention, Caregiver SOS includes 6, 1-hour telephonic sessions with a care manager. Usual care will consist of 1 telephonic session with a care manager. Primary and secondary outcomes will be pre-post change in CG distress and work functioning, respectively. Additional CG and CR outcomes (i.e., physical mental and interpersonal functioning) also will be measured and analyzed. CRs' VA health utilization data will be extracted from clinical patient records and non-VA health utilization data will be collected via CG self-report. Intent to treat analysis using mixed effects models will be used to test the study hypotheses. The investigators anticipate that CGs in the intervention arm will show significantly greater improvements in outcomes compared to those in usual care.

ELIGIBILITY:
Inclusion Criteria:

* Veteran receives care at the Corporal Michael J. Crescenz VA Medical Center (CMCVAMC), VA Western New York Healthcare System (VAWNYHS), or affiliated community-based outpatient clinics
* Veteran and CG are 18 years of age or older
* Veteran and CG are community dwelling
* Veteran has a confirmed diagnosis of depressive disorder, generalized anxiety disorder, PTSD, and/or TBI (per medical chart/provider report)
* CG is a relative or significant other who endorses that s/he assists the Veteran care recipient (CR) with two or more instrumental activities of daily living (IADLs). IADLS include:

  * housework
  * managing finances
  * arranging/providing transportation (e.g., to medical appointments and community services)
  * grocery shopping
  * preparing meals
  * health management and maintenance (e.g., giving medications, minimizing exposure and response to stress triggers)
  * arranging for and/or supervising the delivery of services for assistance with everyday activities
* CG is employed
* CG screens positive for at least mild-moderate distress
* CG screens positive for at least moderate work role difficulty due to caregiving
* CG is willing and able to provide informed consent

Exclusion Criteria:

* CG cognitive, hearing, visual, or other physical impairments leading to difficulty with informed consent process, assessment, or participation in intervention visits
* CG unable to speak or read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy W Helstrom, PhD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA; Laura O Wray, PhD, Principal Investigator — VA Western New York Healthcare System, Buffalo, NY
Locations (2):
- United States (2):
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 300 participants were approved; 199 were recruited. The difference between the actual and targeted sample sizes are due to the multiple changes in staffing as well as the COVID pandemic that stalled initial recruitment.
Groups:
- Caregiver SOS: SOS care is brief, telephonic care (6 one-hour sessions over 3-4 months) tailored to the CG's needs, preferences, and priorities. SOS care addresses both work and caregiving-related stress. The five pillars of behavior change in SOS care are: 1) knowledge of work and CG stress; 2) stress management skills and abilities; 3) supports and resources; 4) confidence and motivation to modify stress; and 5) work and CG-focused problem-solving skills. The pillars are addressed through seven modules. In six sessions, the CM will cover each module at least once. SOS care involves an ongoing process of formulating self-management goals and action plans and preparing CGs to succeed in implementing them. CMs will educate CGs about stress. CMs introduce strategies for self-managing stress and design experiments to test these strategies. Progress is monitored to identify strategies that effectively achieve self management goals.
  CG-SOS care is brief, telephonic care tailored to the CG's needs, preferences, and priorities. SOS care addresses both work and caregiving stress. CG:SOS involves: 1) knowledge of work and CG stress; 2) stress management skills and abilities; 3) supports and resources; 4) confidence and motivation to modify stress; and 5) work and CG-focused problem-solving skills. The pillars are addressed through seven modules. In six sessions, the CM will cover each module at least once. succeed in implementing them. CMs will educate CGs about stress.
Period: Overall Study
Arm/Group | Caregiver SOS | Usual Care
Started | 99 | 100
Completed | 45 | 34
Not Completed | 54 | 66
Not completed — Lost to Follow-up | 54 | 66

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caregiver SOS | Usual Care | Total
Number analyzed (Participants) | 99 | 100 | 199
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 47.89 (11.76) | 46.6 (11.77) | 47.6 (11.77)
Sex: Female, Male [Count of Participants; unit: Participants] — Self-identification of male, female, other category. Population: Gender item skipped by participants.
  Participants
    number analyzed (Participants) | 87 | 94 | 181
    Female | 80 | 88 | 168
    Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 18 | 37
  White | 61 | 80 | 141
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: 10-item Kessler Psychological Distress Scale (K10)
Description: Global measure of psychological distress; scores range from 10-50, with higher scores indicating worse outcomes (higher levels of distress)
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver SOS | Usual Care
Number analyzed (Participants) | 43 | 48
score on a scale | 23.38 (7.56) | 23.79 (8.03)
Statistical Analysis 1: Comparison: Caregiver SOS vs Usual Care; There were no statistical differences between the two treatment groups (chi-square=0.43, p=0.513); Test type: Superiority; p = 0.513, Chi-squared

2. Primary Outcome: Caregiver Work Limitations Questionnaire (C-WLQ) - Mental
Description: 25-item measure capturing the extent to which caregiving has impacted work performance and productivity; scores range from 0-100%, with higher scores indicating worse outcomes (greater work difficulty)
  The C-WLQ Mental Subscale has scores ranging from 0-100%
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver SOS | Usual Care
Number analyzed (Participants) | 43 | 48
units on a scale | 62.15 (21.18) | 59.71 (19.79)
Statistical Analysis 1: Comparison: Caregiver SOS vs Usual Care; Test type: Superiority; p = .184, Mixed Models Analysis

3. Primary Outcome: Caregiver Work Limitations Questionnaire (C-WLQ) - Physical
Description: as for outcome 2
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver SOS | Usual Care
Number analyzed (Participants) | 43 | 48
units on a scale | 30.38 (31.65) | 30.84 (29.09)
Statistical Analysis 1: Comparison: Caregiver SOS vs Usual Care; Test type: Superiority; p = 0.525, Chi-squared

4. Primary Outcome: Caregiver Work Limitations Questionnaire (C-WLQ) - Time
Description: as for outcome 2
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver SOS | Usual Care
Number analyzed (Participants) | 43 | 48
units on a scale | 63.06 (23.9) | 62.41 (23.79)
Statistical Analysis 1: Comparison: Caregiver SOS vs Usual Care; Test type: Superiority; p = 0.723, Chi-squared

5. Primary Outcome: Caregiver Work Limitations Questionnaire (C-WLQ) - Output
Description: as for outcome 2
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver SOS | Usual Care
Number analyzed (Participants) | 43 | 48
units on a scale | 67.12 (25.06) | 65.34 (22.66)
Statistical Analysis 1: Comparison: Caregiver SOS vs Usual Care; Test type: Superiority; p = 0.569, Chi-squared

ADVERSE EVENTS:
Time Frame: Data were collected over the course of 3 years (2020-2023)
Arm/Group | Caregiver SOS | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/100
Other Adverse Events (participants affected / at risk) | 0/99 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT04337021/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT04337021/ICF_002.pdf